CLINICAL TRIAL: NCT04611152
Title: A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared With Intravitreal Aflibercept in Participants With Visual Impairment Secondary to Treatment-naïve Diabetic Macular Edema (DME)
Brief Title: A Trial to Evaluate the Efficacy, Durability, and Safety of KSI-301 Compared to Aflibercept in Participants With Diabetic Macular Edema (DME)
Acronym: GLEAM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet primary endpoint
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P104; 2020-001062-11 (EudraCT Number)
Record Dates: First submitted 2020-10-19; First posted 2020-11-02 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Kodiak; Vascular endothelial growth factor; Anti-VEGF; VEGF; Antibody biopolymer conjugate; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, low; Aflibercept; Eylea; Diabetes mellitus; Diabetes; Diabetic retinopathy; Diabetic macular edema; Macular edema; KSI-301
MeSH Terms: conditions — Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low; Diabetes Mellitus; Diabetic Retinopathy; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two treatment arms: KSI-301 or aflibercept.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For masking purposes, sham injections will be administered at every monthly visit if an active treatment is not administered. To preserve masking, two investigators are required for this study. The masked Investigator will be responsible for the examinations and safety assessments. The unmasked Investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 (Arm A) (Experimental): Intravitreal injection of KSI-301 (5 mg) once every 4 weeks for 3 monthly doses followed by an individualized dosing regimen (every 8 to 24 weeks) via intravitreal injection from Week 16 to Week 100.
  Interventions: Drug: KSI-301; Other: Sham Procedure
- Aflibercept (Arm B) (Active Comparator): Intravitreal injection of aflibercept (2 mg) once every 4 weeks for 5 monthly doses followed by aflibercept (2 mg) once every 8 weeks via intravitreal injection from Week 24 to 100.
  Interventions: Drug: Aflibercept; Other: Sham Procedure

INTERVENTIONS:
Drug: KSI-301 — Intravitreal Injection
  Arms: KSI-301 (Arm A)
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept (Arm B)
Other: Sham Procedure — The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This Phase 3 study will evaluate the efficacy, durability, and safety of KSI-301 compared to aflibercept in participants with treatment-naïve DME.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, double-masked, two-arm, multi-center non-inferiority study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in participants with treatment-naïve DME.

The primary endpoint will be assessed at Year 1; additional secondary endpoints for efficacy will be assessed at Years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Treatment-naïve diabetic macular edema, with vision loss and center involvement (if present) diagnosed within 9 months of screening.
3. BCVA ETDRS letter score between 78 and 25 (-20/25 to 20/320 Snellen equivalent), inclusive, in the Study Eye.
4. CST of ≥ 320 microns on SD-OCT (Heidelberg Spectralis or equivalent on other OCT instruments) as determined by the Reading Center.
5. Decrease in vision determined by the Investigator to be primarily the result of DME.
6. Type 1 or Type 2 diabetes mellitus and a HbA1c of ≤12%.
7. Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

1. Macular edema in the Study Eye considered to be secondary to a cause other than DME.
2. Active iris or angle neovascularization or neovascular glaucoma in the Study Eye.
3. High-risk proliferative diabetic retinopathy characteristics in the Study Eye.
4. History of Pan-retinal Photocoagulation (PRP) laser in the Study Eye within 3 months of screening.
5. Tractional retinal detachment in the Study Eye.
6. Active retinal disease other than the condition under investigation in the Study Eye.
7. Any history or evidence of a concurrent ocular condition present, that in the opinion of the Investigator could require either medical or surgical intervention or affect macular edema or alter visual acuity during the study (e.g., vitreomacular traction, epiretinal membrane).
8. Active or suspected ocular or periocular infection or inflammation in either eye at Day 1.
9. Any prior use of an approved or investigational treatment for DME in the Study Eye (e.g., anti-VEGF, intraocular or periocular steroids, macular laser photocoagulation).
10. Women who are pregnant or lactating or intending to become pregnant during the study.
11. Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg or diastolic value ≥100 mmHg while at rest.
12. Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
13. History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
14. Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (75):
- United States (48):
  - UCSD Jacobs Retina Center, La Jolla, California
  - Retina Consultants of Southern California, Redlands, California
  - California Retina Consultants, Santa Maria, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Colorado Retina Associates PC, Lakewood, Colorado
  - Conneticut Eye Consultants, Danbury, Connecticut
  - Retina Group of Florida, Boca Raton, Florida
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Vitreo Retinal Associates, Gainesville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Springfield Clinic LLP, Springfield, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates PA, Lenexa, Kansas
  - Vitreo Retinal Consultants and Surgeons, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - The Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Retina Northwest, Portland, Oregon
  - Cascade Medical Research Institute, Springfield, Oregon
  - MidAtlantic Retina, Philadelphia, Pennsylvania
  - Retina Research of Beaufort, Beaufort, South Carolina
  - Charleston Neuroscience Institute - West Ashley, Charleston, South Carolina
  - Pametto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Star Retina, Burleson, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Retina Consultants of San Antonio, San Antonio, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye, Spokane, Washington
- Germany (5):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Dietrich Bonhoeffer Klinikum Neubrandenburg, Neubrandenburg, Mecklenburg-Vorpommern
  - St. Elisabeth Krankenhaus, Cologne, North Rhine-Westphalia
  - St Franziskus Hospital, Münster, North Rhine-Westphalia
- Hungary (2):
  - Jahn Ferenc Dél-Pesti Kórház és Rendelointézet, Budapest
  - Ganglion Medical Center, Pécs
- Fondazione PTV Policlinico Tor Vergata, Roma, Italy
- Latvia (4):
  - Signes Ozolinas Doctor Praxis In Ophthalmology, Jelgava
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga Eastern Clinical University Hospital Clinic Bikernieki, Riga
  - Latvian American Eye Center, Riga
- Emanuelli Research & Development Center LLC, Arecibo, Puerto Rico
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - Uvea Klinika, S.R.O., Martin
  - Nemocnica s poliklinikou Trebisov a.s. Ocne oddelenie - jednonova zdravotna starostlivost, Trebišov
  - Fakultna nemocnica Trencin, Trencín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Spain (8):
  - Hospital dos de Maig, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari General de Catalunya - Grupo Quironsalud, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 75 medical centers between September 2020 and February 2022. The first participant was enrolled on 30 September 2020 and the last on 16 February 2022.
Pre-assignment Details: Of 670 screened participants, 460 met eligibility criteria and were randomized to treatment. Each participant contributed only one study eye to this study.
Period: Overall Study
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Started | 230 | 230
Completed (Completed is defined as participants who completed treatment through Week 64.) | 204 | 211
Not Completed | 26 | 19
Not completed — Adverse Event | 9 | 8
Not completed — Non-compliance with study schedule | 1 | 3
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 11 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set defined as all randomized subjects who received any study treatment (KSI-301 or aflibercept). Subjects will be analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B) | Total
Number analyzed (Participants) | 230 | 230 | 460
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 136 | 274
  >=65 years | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9.73) | 61.2 (10.61) | 61.6 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 87 | 167
  Male | 150 | 143 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 32 | 69
  Not Hispanic or Latino | 193 | 198 | 391
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 21 | 21 | 42
  White | 204 | 200 | 404
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Geographic Region [Count of Participants; unit: Participants]
  North America | 177 | 176 | 353
  Rest of World | 53 | 54 | 107
BCVA in the Study Eye, Letters [Mean (Standard Deviation); unit: Letters] | 66.4 (9.78) | 66.6 (9.60) | 66.5 (9.68)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in BCVA
Description: Mean change in best-corrected visual acuity (BCVA) from baseline to the average of Weeks 60 and 64 (using Early Treatment Diabetic Retinopathy Study (ETDRS) Letters). Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Day 1 to Week 64
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 230 | 230
ETDRS Letters | 5.6 (0.83) | 9.5 (0.85)
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable true difference between KSI-301 and aflibercept participants to be considered non-inferior is 4.5 ETDRS letters, i.e. the non-inferiority margin; p = 0.4162, Mixed Models Analysis; MMRM model with treatment, visit, treatment by visit interaction, randomization stratification factors, and continuous baseline BCVA and OCT CST; Adjusted mean difference = -3.8, 95.04% CI 2-sided [-5.47 to -2.17], Standard Error of Mean 0.84

2. Secondary Outcome: Percentage of Patients With a ≥ 2-step Worsening on the ETDRS DRSS in Studies KS301P104 and KS301P105 Combined
Description: Percentage of patients with a ≥ 2-step worsening on the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 52 using last observation carried forward (LOCF) in Studies KS301P104 and KS301P105 combined. The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 52
Population: All randomized subjects in Studies KS301P104 and KS301P105 who received any study treatment (KSI-301 or aflibercept) with evaluable results at baseline and evaluable results on or prior to Week 52. The population for studies KS301P104 and KS301P105 are identical in terms of treatment indication and inclusion/exclusion criteria. Please refer to NCT04603937 to review demographics, other study details and adverse events for participants in KS301P105 study.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 433 | 437
Participants | 6 | 3
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable non-inferiority margin between KSI-301 and aflibercept subjects is 10% to be considered non-inferior, i.e. the "non-inferiority margin" is 10%; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haentzel test stratified by study identifier and randomization stratification variables; Difference of weighted percentages = 0.6, 95.04% CI 2-sided [-0.7 to 2] — Weighted percentages are based on weighted average of observed estimates across strata using CMH weights. The CI are based on the normal approximation to the binomial proportions

3. Secondary Outcome: Percentage of Patients With a ≥ 2-step Worsening on the ETDRS DRSS in Study KS301P104
Description: Percentage of patients with a ≥ 2-step worsening on the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 52 using last observation carried forward (LOCF) in Study KS301P104. The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 52
Population: All randomized subjects who received any study treatment (KSI-301 or aflibercept) with evaluable results at baseline and evaluable results on or prior to Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 215 | 219
Participants | 0 | 0
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference of weighted percentages = 0, 95.04% CI 2-sided [0 to 0] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Patients in the KSI-301 Arm on a Q8W, Q12W, Q16W, Q20W, or Q24W Treatment Interval
Description: Percentage of patients in the KSI-301 arm on a Q8W, Q12W, Q16W, Q20W, or Q24W treatment interval at the primary endpoint. Analyses include KSI-301 patients who completed a treatment interval from Week 56 onwards.
Time Frame: Week 56
Population: Analyses include KSI-301 patients who completed a treatment interval from Week 56 onwards.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A)
Number analyzed (Participants) | 208
Participants
  Number of participants on the KSI-301 Q8W | 61
  Number of participants on the KSI-301 Q12W | 21
  Number of participants on the KSI-301 Q16W | 19
  Number of participants on the KSI-301 Q20W | 8
  Number of participants on the KSI-301 Q24W | 99

5. Secondary Outcome: Mean Number of Intravitreal Injections
Description: Mean number of intravitreal injections from Day 1 to Week 60
Time Frame: Day 1 to Week 60
Population: Safety Analysis Set includes all patients who received any study treatment (KSI-301 or aflibercept).
  Patients will be analyzed according to the study treatment they actually received.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 230 | 230
injections | 5.9 (1.71) | 9.2 (1.46)

6. Secondary Outcome: Mean Change in OCT CST
Description: Mean change in Optical Coherence Tomography (OCT) central subfield retinal thickness (CST) from baseline to the average of Weeks 60 and 64
Time Frame: Day 1 to Week 64
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 230 | 230
Microns | -140.4 (132.7) | -158.5 (121.75)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported through Week 64 or Early Termination (ET) if occurred before Week 64.
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
All-Cause Mortality (participants affected / at risk) | 5/230 | 5/230
Serious Adverse Events (participants affected / at risk) | 61/230 | 51/230
Other Adverse Events (participants affected / at risk) | 126/230 | 121/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=230) | Aflibercept (Arm B) (N=230)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3)
Coronary artery disease (Cardiac disorders) | 4 (4) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 3 (5) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2)
Osteomyelitis (Infections and infestations) | 4 (4) | 3 (4)
Cellulitis (Infections and infestations) | 4 (5) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Gangrene (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Diabetic gangrene (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis - Study Eye (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical observation (Investigations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endocrine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6)
Hypertensive urgency (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=230) | Aflibercept (Arm B) (N=230)
Cataract - Study Eye (Eye disorders) | 35 (38) | 17 (17)
Diabetic retinal oedema - Fellow Eye (Eye disorders) | 19 (19) | 21 (22)
Conjunctival haemorrhage - Study Eye (Eye disorders) | 18 (21) | 15 (21)
Cataract - Fellow Eye (Eye disorders) | 15 (15) | 12 (12)
Dry eye - Study Eye (Eye disorders) | 13 (15) | 10 (11)
COVID-19 (Infections and infestations) | 42 (45) | 33 (36)
Nasopharyngitis (Infections and infestations) | 8 (8) | 17 (18)
Diabetes mellitus (Metabolism and nutrition disorders) | 19 (19) | 17 (18)
Chronic kidney disease (Renal and urinary disorders) | 8 (8) | 14 (14)
Hypertension (Vascular disorders) | 30 (33) | 31 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT04611152/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04611152/SAP_001.pdf